CLINICAL TRIAL: NCT01057927
Title: Parallel Group, Randomised, Placebo Controlled, Double Blind Oral Assessment of OC000459 Dosed Twice Daily for 28 Days in Asthmatic Subjects
Brief Title: Safety and Efficacy Study of OC000459 Dosed Twice Daily for 28 Days in Asthmatic Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oxagen Ltd (Industry)
Responsible Party: Dr C Mike Perkins, Oxagen Ltd
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OC000459/006/06
Record Dates: First submitted 2010-01-25; First posted 2010-01-28 (Estimated); Last update posted 2010-01-28 (Estimated); Status verified 2010-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — (5-fluoro-2-methyl-3-quinolin-2-ylmethylindo-1-yl)acetic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OC000459 (Experimental)
  Interventions: Drug: OC000459
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OC000459 — OC000459 capsules 2x100mg BID for 28 days
  Arms: OC000459
Drug: Placebo — Placebo capsules to match OC000459 100mg capsules, 2 tablets BID
  Arms: Placebo

SUMMARY:
The purpose of the study is to investigate the clinical effects of multiple (28 day) twice-daily doses of OC000459 in comparison to placebo on clinic lung function (FEV1) in mild to moderate asthmatics with an FEV1 of 60-80% of predicted and requiring only short acting inhaled B2-adrenergic agonists for symptomatic control.

ELIGIBILITY:
Inclusion Criteria At Screening:

* Male or female asthmatics, any racial group. Females of childbearing potential must practise two forms of contraception
* Non smokers
* Mild to moderate asthmatics according to GINA guidelines for at least 12 months.
* History of asthma symptoms increasing in response to external allergens.
* Testing positive on skin prick test to an allergen associated with the subject's asthma

Exclusion Criteria:

* Use of inhaled or local corticosteroids in the period from 28 days prior to screening.
* Receipt of prescribed or over the counter medication within 14 days of the first study day.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2007-01; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Forced expiratory volume in one second (FEV1) | 28 days

SECONDARY OUTCOMES:
Clinic peak expiratory flow, diary peak expiratory flow, diary asthma symptoms, diary salbutamol use, Asthma Quality of Life Questionnaire (AQLQ(S)) | 28 days
Sputum eosinophilia (subset of patients) and serum IgE | 28 days
Safety and tolerability assessed by adverse events, chest examination, concomitant medication and laboratory safety parameters | 28 days

CONTACTS AND LOCATIONS:
Locations (16):
- Russia (16):
  - Research Institute of Pulmonology, Moscow
  - Burdenko Main Military Hospital, Moscow
  - City Hospital #23, Moscow
  - City Hospital #7, Moscow
  - Vishnevsky Central Military Hospital #3, Moscow
  - Leningrad Regional Hospital, Saint Petersbrug
  - St George City Hospital, Saint Petersbrug
  - St Petersburg Medical Academy of Postgraduate Education, Saint Petersburg
  - St Petersburg Medical Academy, Saint Petersburg
  - Outpatient Clinic #94, Saint Petersburg
  - St Petersbrug Hospital of the Russian Academy of Science, Saint Petersburg
  - Russian Center of Emergency and Radiology Medicine, Saint Petersburg
  - St Petersburg State Pediatrics Academy, Saint Petersburg
  - Central Medical Unit #122, Saint Petersburg
  - St George City Hospital, Saint Petersburg
  - Sverdlovsk Regional Hospital #1, Yekaterinburg

REFERENCES:
- [Derived] Barnes N, Pavord I, Chuchalin A, Bell J, Hunter M, Lewis T, Parker D, Payton M, Collins LP, Pettipher R, Steiner J, Perkins CM. A randomized, double-blind, placebo-controlled study of the CRTH2 antagonist OC000459 in moderate persistent asthma. Clin Exp Allergy. 2012 Jan;42(1):38-48. doi: 10.1111/j.1365-2222.2011.03813.x. Epub 2011 Jul 15. PMID 21762224